CLINICAL TRIAL: NCT05371106
Title: Maternal and Newborn Exposure to Mycotoxins in Israel and the Association to Baby's Development in First Months of Life
Brief Title: Mycotoxins in Mothers Milk in Israel
Status: Recruiting | Type: Observational
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 224-20-ASF
Record Dates: First submitted 2022-04-25; First posted 2022-05-12 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Breastfeeding
Keywords: mycotoxins
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — milk
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- breastfeeding mothers: pregnant women after week 37 intending to nurse or nursing mothers of infants aged 1-12 months
  Interventions: Other: exposure to mycotoxins

INTERVENTIONS:
Other: exposure to mycotoxins — self-report eating questionnaire

SUMMARY:
Some plant pathogen fungi may develop in grains, nuts and dry foodstuff during their storage. They secrete toxins which are very resistant and persistent.

The toxins enter the human body through the food. Women eating without their knowledge spoiled food absorb the toxin which is conveyed into their milk. In the same way, meat and dairy products can be contaminated with mycotoxins.

Toxins and their metabolites can have negative effects on pregnant women and on the fetus or infant health.

The main purpose of this trial is to assess the presence of toxins in mothers's milk.

DETAILED DESCRIPTION:
Fungi from the genus Aspergillus, Penicillium, Fusarium and Alternaria can synthesize toxins. These may be carcinogenic, immunotoxic or endocrine disruptors.

In this trial, Zearalenone, Deoxynivalenol, T-2 toxin, Fumonisin B1, Fumonisin B2, Aflatoxin M1, Aflatoxin B1, Aflatoxin B2, Aflatoxin G1, Aflatoxin G2, Ochratoxin A, HT-2 toxin, De-epoxy-deoxynivalanol presence and quantity will be assessed in mother's milk.

Another purpose is to try to pinpoint at the source(s) of contamination.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 and above.
* Pregnant women after week 37 intending to breastfeed.
* Women breastfeeding.

Exclusion Criteria:

* Women taking drugs which influence milk production.
* Women taking drugs contraindicated during breastfeeding.
* Women not staying in Israel during third trimester or in the months after birth for a long period of time.
* Women not wanting/able to fill up the questionnaires.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: pregnant women after week 37 intending to nurse or nursing mothers of infants aged 1-12 months
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Mycotoxins in breastmilk | approx. 6 months after recruitment
  To measure mycotoxins and mycotoxins metabolites levels in breast milk

SECONDARY OUTCOMES:
Source of contamination | approx. one year after recruitment
  To evaluate the source of the contamination by correlation to food intake and life habits questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Elkana Kohn, Ph.D., Principal Investigator — Shamir (Assaf Harofeh) Medical Center
Locations (1):
- Assaf Harofeh Medical Center, Ẕerifin, Israel

IPD SHARING:
Plan to Share IPD: Yes
The study protocol will be shared with researchers
Supporting Information: Study Protocol
Time Frame: starting 6 months after publication
Access Criteria: interested colleagues

REFERENCES:
- [Background] Wild CP, Gong YY. Mycotoxins and human disease: a largely ignored global health issue. Carcinogenesis. 2010 Jan;31(1):71-82. doi: 10.1093/carcin/bgp264. Epub 2009 Oct 29. PMID 19875698
- [Background] Tesfamariam K, De Boevre M, Kolsteren P, Belachew T, Mesfin A, De Saeger S, Lachat C. Dietary mycotoxins exposure and child growth, immune system, morbidity, and mortality: a systematic literature review. Crit Rev Food Sci Nutr. 2020;60(19):3321-3341. doi: 10.1080/10408398.2019.1685455. Epub 2019 Nov 6. PMID 31694387
- [Background] Warth B, Braun D, Ezekiel CN, Turner PC, Degen GH, Marko D. Biomonitoring of Mycotoxins in Human Breast Milk: Current State and Future Perspectives. Chem Res Toxicol. 2016 Jul 18;29(7):1087-97. doi: 10.1021/acs.chemrestox.6b00125. Epub 2016 Jun 28. PMID 27300310
- [Background] El-Tras WF, El-Kady NN, Tayel AA. Infants exposure to aflatoxin M(1) as a novel foodborne zoonosis. Food Chem Toxicol. 2011 Nov;49(11):2816-9. doi: 10.1016/j.fct.2011.08.008. Epub 2011 Aug 16. PMID 21864634